CLINICAL TRIAL: NCT00852306
Title: A Comparison of Two Freezing Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-265
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Infertility
Keywords: oocyte freezing; vitrification; slow freeze; fertility preservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- slow freeze (Experimental): these recipients will have their first embryo transfer with oocytes frozen via the slow freeze method.
  Interventions: Procedure: oocyte freezing
- vitrification (Experimental): these recipients will have their first attempt at an embryo transfer with oocytes frozen via the vitrification method.
  Interventions: Procedure: oocyte freezing

INTERVENTIONS:
Procedure: oocyte freezing — retrieved oocytes from the donor will be split in half and frozen by both existing egg freezing methods: slow freezing and vitrification. The recipients will then be randomized as to which group of eggs will be thawed out for their first attempt at achieving a pregnancy.

SUMMARY:
The purpose of this study is to determine the best way to freeze eggs in order to preserve the fertility potential of young women.

DETAILED DESCRIPTION:
Human egg freezing is rapidly becoming a vital tool in Assisted Reproductive Technology. Candidates for egg freezing include women without partners who wish to preserve their fertility; cancer patients at risk of losing fertility from chemotherapy; and donor egg recipients. While in the past, egg freezing has not been as successful as embryo freezing in producing live births, recent experience in several centers has demonstrated significant improvement, with pregnancy rates comparable to those achieved with frozen embryos. The purpose of this study is to determine the best method to freeze eggs. We shall be seeking volunteers from the egg donor program, since young, fertile donors represent the best model to study the effect of egg freezing.

We plan to enroll 12 recipients and 6 donors in this study. Each egg donor will go through a stringent screening process (medical, genetic and psychological). Eggs retrieved from all donors will be split in half: one half will be frozen by the slow freeze method, and the other half by vitrification. Each of the six donors will be paired with two recipients; each recipient will be assigned half the total eggs frozen. For each recipient, half of the eggs will come from the slow freeze group and the other half will come from vitrification.

When the recipient's uterine lining is deemed ready (following estrogen treatment and ultrasound monitoring), thawing will be performed on eggs frozen by either the slow freeze or the vitrification method. The thaw process will be randomized between the two types of freezing. One sperm will be injected into each egg that survived the freeze. Fertilization and embryo development will be recorded. Ideally, two embryos will be transferred into the recipient's uterus. Pregnancy will be determined by a blood test and followed by serial blood tests and ultrasound.

The study will determine which freezing method yields better survival and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* donors: women ages 21-32 who wish to donate their eggs; must pass medical, physical and psychological screening.
* recipients: women under the age of 50 who wish to have eggs donated to them through the Donor Egg Program and who aslo pass the medical, physical and psychological screening.

Exclusion Criteria:

* donors: those who do not pass the genetic screening or psychological testing, as described below
* recipients: those who do not pass the screening.

The genetic screening of donors will involve the following:

* All donors will be screened for Cystic Fibrosis, Fragile X and Spinomuscular Atrophy (SMA).
* In addition, donors of Ashkenazi Jewish origin will be screened for Gaucher's disease, Canavan,Tay -Sachs, Familial Dysautonomia, Niemann Pick, Fanconi's Anemia, Bloom and Mucolipidosis Type IV.
* Donors of African-American origin will be screened for Sickle-Cell disease.
* Donors of Asian, Mediterranean, Latino or Hispanic origins will be screened for Thalassemia.

Recipient Screening: A Reproductive Endocrinologist (RE) at the Center will take a detailed history and perform a physical examination on all potential recipients. The RE will assess the health of the potential recipient in order to assess her capacity to carry a pregnancy. Previous IVF cycles, successful or unsuccessful, will have no implication on recipient selection.

The recipient and her partner (if applicable) will meet with the program psychologist. The psychological evaluation is detailed below.

Psychological evaluation: A psychological evaluation will be conducted of the Recipient, her partner (if applicable) and the Donor. The purpose of these evaluations is to determine the suitability of the parties to participate in the Donor Egg Program. Psychological tests will be administered by the Center as part of the evaluation process.

These evaluations may result in a recommendation that one and/or all of the parties not participate in the Donor Egg Program. The psychologist will not be providing any advice or treatment to the Donor or Recipient(s). Nor will the Donor or Recipient(s) be entitled to the results of the Psychologist's evaluation. The Psychologist will provide the results of his/her evaluations to the Center for Human Reproduction.

As with our standard Donor Egg Program practices, there will be an upper age limit of 50 years for all recipients participating in the study.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Achievement of a pregnancy, as determined by a fetal heartbeat | 2 months

SECONDARY OUTCOMES:
Percentage of eggs that result in blastocyst formation | 1 week
Oocyte survival (the percentage of eggs that survive the freeze-thaw procedure) | 2 days
ICSI fertilization rate (percentage of eggs that fertilize) | 2 days
Incidence rate of embryo formation (percentage of embryos formed/number of eggs fertilized) | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Avner Hershlag, MD, Principal Investigator — Northwell Health; Matthew Cohen, MD, Principal Investigator — Northwell Health; Huai L Feng, PhD, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

REFERENCES:
- [Background] Cohen J, Alikani M, Trowbridge J, Rosenwaks Z. Implantation enhancement by selective assisted hatching using zona drilling of human embryos with poor prognosis. Hum Reprod. 1992 May;7(5):685-91. doi: 10.1093/oxfordjournals.humrep.a137720. PMID 1639990
- [Background] Diaz DG, Rodriguez-Karl MC and Moody JE (2007) Human oocyte cryopreservation: preliminary results of survival, fertilization and cleavage rate of frozen oocyte using a new modified slow-freeze protocol. Fertil Steril 88, Suppl 1:S47.
- [Background] Smith GD, Serafini PC, Fioravanti J, Yadid I, Coslovsky M, Hassun P, Alegretti JR, Motta EL. Prospective randomized comparison of human oocyte cryopreservation with slow-rate freezing or vitrification. Fertil Steril. 2010 Nov;94(6):2088-95. doi: 10.1016/j.fertnstert.2009.12.065. Epub 2010 Feb 19. PMID 20171613
- [Background] Fosas N, Marina F, Torres PJ, Jove I, Martin P, Perez N, Arnedo N, Marina S. The births of five Spanish babies from cryopreserved donated oocytes. Hum Reprod. 2003 Jul;18(7):1417-21. doi: 10.1093/humrep/deg297. PMID 12832365
- [Background] Gook DA, Edgar DH. Human oocyte cryopreservation. Hum Reprod Update. 2007 Nov-Dec;13(6):591-605. doi: 10.1093/humupd/dmm028. Epub 2007 Sep 10. PMID 17846105
- [Background] Hershlag A, Paine T, Kvapil G, Feng H, Napolitano B. In vitro fertilization-intracytoplasmic sperm injection split: an insemination method to prevent fertilization failure. Fertil Steril. 2002 Feb;77(2):229-32. doi: 10.1016/s0015-0282(01)02978-8. PMID 11821076
- [Background] Jain JK, Paulson RJ. Oocyte cryopreservation. Fertil Steril. 2006 Oct;86(4 Suppl):1037-46. doi: 10.1016/j.fertnstert.2006.07.1478. PMID 17008147
- [Background] Kumayama M and Kato O (2000a) Successful vitrification of human oocytes. Fertil Steril 74, Suppl 3:S49.
- [Background] Kumayama M and Kato O (2000b) All-round vitrification method for human oocytes and embryos. J Asst Reprod Gen 17:447.
- [Background] Kuzan FB and Quinn P (1988) Cryopreservation of mammalian embryos IN in vitro fertilization and embryo transfer: a manual of basic techniques. Plenum Press, New York.
- [Background] Li Y, Feng HL, Cao YJ, Zheng GJ, Yang Y, Mullen S, Critser JK, Chen ZJ. Confocal microscopic analysis of the spindle and chromosome configurations of human oocytes matured in vitro. Fertil Steril. 2006 Apr;85(4):827-32. doi: 10.1016/j.fertnstert.2005.06.064. PMID 16580356
- [Background] Nagy ZP, Chang CC, Shapiro DB, Bernal DP, Elsner CW, Mitchell-Leef D, Toledo AA, Kort HI. Clinical evaluation of the efficiency of an oocyte donation program using egg cryo-banking. Fertil Steril. 2009 Aug;92(2):520-6. doi: 10.1016/j.fertnstert.2008.06.005. Epub 2008 Aug 9. PMID 18692830
- [Background] Oktay K, Cil AP, Bang H. Efficiency of oocyte cryopreservation: a meta-analysis. Fertil Steril. 2006 Jul;86(1):70-80. doi: 10.1016/j.fertnstert.2006.03.017. PMID 16818031
- [Background] Palermo G, Joris H, Devroey P, Van Steirteghem AC. Pregnancies after intracytoplasmic injection of single spermatozoon into an oocyte. Lancet. 1992 Jul 4;340(8810):17-8. doi: 10.1016/0140-6736(92)92425-f. PMID 1351601
- [Background] Paynter SJ. Current status of the cryopreservation of human unfertilized oocytes. Hum Reprod Update. 2000 Sep-Oct;6(5):449-56. doi: 10.1093/humupd/6.5.449. PMID 11045876
- [Background] Porcu E, Venturoli S. Progress with oocyte cryopreservation. Curr Opin Obstet Gynecol. 2006 Jun;18(3):273-9. doi: 10.1097/01.gco.0000193015.96275.2d. PMID 16735826
- [Background] Tucker M, Wright G, Morton P, Shanguo L, Massey J, Kort H. Preliminary experience with human oocyte cryopreservation using 1,2-propanediol and sucrose. Hum Reprod. 1996 Jul;11(7):1513-5. doi: 10.1093/oxfordjournals.humrep.a019428. PMID 8671495
- [Background] Wolf DP (1991) ProH2 freeze/thaw protocol for human embryos IN OHSU procedure manual.
- [Background] Wu J, Zhang L, Wang X. In vitro maturation, fertilization and embryo development after ultrarapid freezing of immature human oocytes. Reproduction. 2001 Mar;121(3):389-93. doi: 10.1530/rep.0.1210389. PMID 11226064
- [Background] Yoon TK, Kim TJ, Park SE, Hong SW, Ko JJ, Chung HM, Cha KY. Live births after vitrification of oocytes in a stimulated in vitro fertilization-embryo transfer program. Fertil Steril. 2003 Jun;79(6):1323-6. doi: 10.1016/s0015-0282(03)00258-9. PMID 12798878
- [Background] Yoon TK, Chung HM, Lim JM, Han SY, Ko JJ, Cha KY. Pregnancy and delivery of healthy infants developed from vitrified oocytes in a stimulated in vitro fertilization-embryo transfer program. Fertil Steril. 2000 Jul;74(1):180-1. doi: 10.1016/s0015-0282(00)00572-0. No abstract available. PMID 10899519